CLINICAL TRIAL: NCT06081608
Title: Acute Kidney Injury Among Pediatric Cancer Patients At South Egypt Cancer Institute
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Amir Fathy Riad, resident doctor, Assiut University
Other Study IDs: 639
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: To Determine the Cumulative Incidence of AKI Using KDIGO Criteria in Pediatric Patients With Malignancy in South Egypt Cancer Institute (SECI)
MeSH Terms: interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

INTERVENTIONS:
Diagnostic Test: kidney function test — blood sample for kidney function test

SUMMARY:
Cancer is the second most frequent cause of premature death in children. The incidence of pediatric cancer varies by region and country, but it is generally considered rare with an estimated 300,000 new cases diagnosed worldwide. Acute kidney injury in pediatric cancer patients refers to the sudden and often temporary loss of renal function, which can lead to a variety of complications if not treated correctly.

DETAILED DESCRIPTION:
* Primary: To determine the cumulative incidence of AKI using KDIGO criteria in pediatric patients with malignancy in South Egypt Cancer Institute (SECI)
* Secondary:

  1. Incidence of Hospital-acquired and community-acquired AKI
  2. Asses the risk factors of the incidence of AKI
  3. To determine in-hospital outcome (time to in-hospital death, length of hospital stay, and time to kidney recovery) of AKI.

This is a prospective study that will be carried out in the Paediatric Oncology and Haematological Malignancies Department including patients diagnosed with malignant tumours and hospitalized from 1st April 2023 for one year duration.

ELIGIBILITY:
Inclusion Criteria:

* • Children of both sexes (aged from 1 month to 18 years at diagnosis)

  * Patients with either hematological malignancies or solid tumors admitted to the Paediatric Oncology and Haematological Malignancies Department

Exclusion Criteria:

* Children who had an unconfirmed cancer diagnosis.
* Children more than 18 years at diagnosis.
* Children with preexisting chronic kidney disease (CKD) that defined as the presence of structural or functional kidney damage that persist over minimum of three month
* The patient underwent hematopoietic stem cell transplantation. Patients with 1 s.Cr level.
* Patient underwent renal transplant.

Ages: 30 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: •Children of both sexes (aged from 1 month to 18 years at diagnosis)
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine the cumulative incidence of AKI using KDIGO criteria in pediatric patients with malignancy in South Egypt Cancer Institute (SECI) | from November 2023 till November 2024

IPD SHARING:
Plan to Share IPD: Undecided